CLINICAL TRIAL: NCT00480285
Title: A Prospective Randomized Trial Comparing Laparoscopic Nissen Against Anterior Partial Fundoplication in Treating Gastroesophageal Reflux Disease Among Chinese Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE2006.287-T
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Laparoscopic Nissen Fundoplication; Laparoscopic anterior partial fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic Nissen Fundoplication
Procedure: Laparoscopic anterior partial fundoplication

SUMMARY:
The aim of this study is to compare the effectiveness of laparoscopic Nissen against anterior partial fundoplication in the control of gastroesophageal reflux disease among Chinese patients

Study hypothesis Laparoscopic Nissen is comparable to anterior partial fundoplication in the control of gastroesophageal reflux disease

DETAILED DESCRIPTION:
The incidence of gastroesophageal reflux disease (GERD) is rising among Asian population. A recent systematic review showed among Chinese population, the prevalence of GERD can be up to 5% (2). Currently, the standard treatment for GERD is acid suppression using proton pump inhibitors (PPI) which can achieve a symptomatic relief of more than 90%. However, more than 50% of patients with GERD will required long term PPI. As the usual occurrence of GERD is at the age of 40 to 50, the need of long term PPI among these young adults renders them playing a sick role for a long period of time. This imposed a major impact on these patients' quality of life, and a significant medical expenditure to the society.

Since Rudolf Nissen first reported the use of fundoplication as a treatment of gastroesophageal reflux disease in 1956, there has been a development in variety of different fundoplication. It can be classified into a complete or partial wrapping at the lower esophageal sphincter around the esophago-gastric junction (EGJ). From the results of numerous randomized studies, Fundoplication is considered as an alternative to long term proton pump inhibitors. Recent controversies abound upon the use of partial or complete fundoplication. Several randomized studies reported that a partial fundoplication can reduce the incidence of post-operative dysphagia. However, this benefit is off-set by an increase in the incidence of recurrence. From our retrospective review on 28 patients treated by laparoscopic fundoplication, the recurrence of GERD is significantly higher in patients treated with partial compared to a complete fundoplication. The effectiveness of partial against complete Nissen fundoplication in control of reflux among Chinese patients is still unknown. Our study aimed to compare Laparoscopic Nissen fundoplication against Anterior partial on the control of gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 and < 70
* Gastroesophageal reflux disease (GERD) as evidence by

  1. Typical symptoms including heartburn &/or acid regurgitation &/or acid in throat
  2. Good response to PPI therapy

     * Defined as a complete cessation of GERD symptoms (as above) with 4 weeks of high dose PPI
     * PPI - standardized to Esomeprazole 40mg daily
  3. Not able to wean off PPI to on-demand regimen

Exclusion Criteria:

* Achalasia
* Moribund patients
* Pregnancy
* Previous gastrectomy / esophagectomy
* Informed consent not available
* Non-Chinese ethnic group
* Patients with hiatus hernia > 3cm (measured by endoscopy & / or manometry)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of gastroesophageal reflux disease that required medication therapy | 5 years

SECONDARY OUTCOMES:
1. Dysphagia - measured by the 4-point Likert scale (0 - no dysphagia,1 - mild dysphagia, 2 - moderate dysphagia, 3 - severe dysphagia)
2. Ability to bloat / belch
3. Overall Satisfaction - (0 - Very satisfactory, 1 - Good, 2 - no comment, 3 - Unsatisfactory)
4. Quality of life score - measure by SF36 before operation, 6 months and 12 months after operation
5. GERD related QoL assessment
6. Perioperative outcomes - hospital stay, operative time, morbidity, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Chiu, FRCSEd, Principal Investigator — Surgery, Institute of Digestive Disease, The Chinese University of Hong Kong
Locations (1):
- Philip Chiu, Hong Kong, Hong Kong